CLINICAL TRIAL: NCT05184075
Title: A Randomized Controlled Trial to Investigate the Ideal Sequence of Hybrid Coronary Revascularization with Endoscopic Coronary Revascularization
Brief Title: The Ideal Sequence of Hybrid Coronary Revascularization with Endoscopic Coronary Revascularization
Acronym: HYBRID
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After the passing of the cardiac surgeon, the clinical trial could not be continued.
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: f/2021/085
Record Dates: First submitted 2021-12-20; First posted 2022-01-11 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease
Keywords: Hybrid coronary revascularization; Coronary revascularization
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reverse hybrid coronary revascularization (HCR) (Active Comparator): Patients will undergo reverse hybrid coronary revascularization. Moreover, quality of life is assessed at baseline, 14 days, 30 days, 90 days, 6 months and 1 year.
  Interventions: Procedure: Reverse hybrid coronary revascularization
- Standard hybrid coronary revascularization (HCR) (Active Comparator): Patients will undergo standard hybrid coronary revascularization. Moreover, quality of life is assessed at baseline, 14 days, 30 days, 90 days, 6 months and 1 year.
  Interventions: Procedure: Standard hybrid coronary revascularization

INTERVENTIONS:
Procedure: Standard hybrid coronary revascularization — Patients will undergo endoscopic coronary artery bypass grafting (endo-CABG) within four weeks after the diagnostic coronarography. Furthermore, they will receive a percutaneous coronary intervention (PCI) within four weeks after the endo-CABG.
  Arms: Standard hybrid coronary revascularization (HCR)
Procedure: Reverse hybrid coronary revascularization — Patients will receive a percutaneous coronary intervention (PCI) within four weeks after the diagnostic coronarography. Furthermore, they will undergo the endoscopic coronary artery bypass grafting (endo-CABG) within four weeks after the PCI.
  Arms: Reverse hybrid coronary revascularization (HCR)

SUMMARY:
Hybrid coronary revascularization (HCR), a combination of coronary artery bypass graft surgery (CABG) and percutaneous coronary intervention (PCI), has emerged as an alternative treatment for multivessel coronary artery disease patients. However, the ideal sequence (PCI or CABG) is unclear.

The overall aim of this study is to investigate the best sequence within hybrid coronary revascularization using endoscopic coronary bypass grafting (i.e., first CABG then PCI versus first PCI then CABG)

DETAILED DESCRIPTION:
Hybrid coronary revascularization (HCR) is an emerging approach for multivessel coronary artery disease (MVD) which combines the excellent long-term outcomes of surgery with the early recovery and reduced short-term complications of percutaneous coronary intervention (PCI). However, the best sequence within hybrid coronary revascularization remains unclear. When CABG is performed first (standard HCR), incomplete revascularization can cause acute coronary events in the interim period. On the other hand, when PCI is performed first (reverse HCR), bleeding risks may be higher since CABG should be performed on uninterrupted dual anti-platelet therapy (DAPT). The use of minimally invasive surgery techniques is associated with reduced bleeding because of the less surgical trauma and may offer the opportunity to perform reverse HCR due to the possibility to reduce the risk of bleeding.

The overall aim of this study is to investigate the best sequence within hybrid coronary revascularization using endoscopic coronary bypass grafting (i.e., first CABG then PCI versus first PCI then CABG, figure 1)

ELIGIBILITY:
Inclusion Criteria:

* Multivessel coronary disease, defined as ≥ 50% diameter stenosis by visual estimation in 2 or more of the three major epicardial vessels or major side branches, with at least one or more one stenosis amenable to revascularization with PCI, if the patient cannot be full revascularized by surgery for a specific reason as determined by the Heart Team. Patients with a non-dominant right coronary artery may be included if the left anterior descending artery (LAD) and left circumflex have ≥50% stenosis.
* Age 18-85
* Willing and able to provide informed, written consent

Exclusion Criteria:

* Requirement for other cardiac or non-cardiac surgical procedures (e.g., valve replacement, carotid revascularization)
* Cardiogenic shock and/or need for mechanical/pharmacologic hemodynamic support at the time of randomisation
* Left main coronary artery disease
* Contraindication for dual antiplatelet therapy
* ST-Elevation Myocardial Infarction (STEMI)
* Previous cardiac surgery
* Participation in other interventional clinical trials
* Recent coronary intervention (PCI)
* Ongoing high risk non-ST-segment elevation acute coronary syndrome (ACS)
* Life expectancy < 1 year
* Active bleeding more or equal to BARC 2 at time of randomisation
* Requiring renal replacement therapy
* Undergoing evaluation for organ transplantation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-11-09 (Actual); Study Completion 2024-11-09 (Actual)

PRIMARY OUTCOMES:
30-day net adverse clinical event (NACE) | From the first procedure until 30 days after the second procedure.
  NACE consists of major adverse cardiac and cerebrovascular events (MACCE) and major bleeding unrelated to CABG (Bleeding Academic Research Consortium (BARC) type 3 and 5)
  MACCE consists of:
  * Death from any cause
  * Myocardial infarction
  * Stroke
  * Target lesion revascularisation

SECONDARY OUTCOMES:
Key secondary outcome: 30-day major adverse cardiac and cerebrovascular events (MACCE) | From the first procedure until 30 days after the second procedure
  MACCE consists of:
  * Death from any cause
  * Myocardial infarction
  * Stroke
  * Target lesion revascularisation
Key secondary outcome: 30-day major or clinically relevant non-major bleeding (BARC type 2, 3, 4, 5) | From the first procedure until 30 days after the second procedure
  Major or clinically relevant non-major bleeding is assessed using BARC type 2, 3, 4, and 5.
Key secondary outcome: One-year net adverse clinical event (NACE) | From the first procedure until one year after the second procedure
  NACE consists of major adverse cardiac and cerebrovascular events (MACCE) and major bleeding unrelated to CABG (Bleeding Academic Research Consortium (BARC) type 3 and 5)
  MACCE consists of:
  * Death from any cause
  * Myocardial infarction
  * Stroke
  * Target lesion revascularisation
Key secondary outcome: one-year major adverse cardiac and cerebrovascular events (MACCE) | From the first procedure until one year after the second procedure
  MACCE consists of:
  * Death from any cause
  * Myocardial infarction
  * Stroke
  * Target lesion revascularisation
Key secondary outcome: One-year major or clinically relevant non-major bleeding (BARC type 2, 3, 4, 5) | From the first procedure until one year after the second procedure
  Major or clinically relevant non-major bleeding is assessed using BARC type 2, 3, 4, and 5.
Mortality | From the first procedure until one year after the second procedure
  Both all-cause mortality as the subdivision in cardiovascular death, noncardiovascular death and undetermined cause of death are examined.
Myocardial infarction | From the first procedure until one year after the second procedure
  Mycardial infarction is subdivided into:
  * Periprocedural
  * Spontaneous
Stent thrombosis | From the first procedure until one year after the second procedure
  Stent thrombosis is subdivided into:
  * Definite stent thrombosis
  * Probable stent thrombosis
  * Possible stent thrombosis
Stroke | From the first procedure until one year after the second procedure
  Stroke is subdivided into:
  * Ischemic stroke
  * Hemorrhagic stroke
  * Non-specified stroke
Revascularization | From the first procedure until one year after the second procedure
  Revascularization is subdivided into:
  * Target lesion revascularization (TLR)
  * Target vessel revascularization (TVR)
Graft failure | From the first procedure until one year after the second procedure
  Graft failure describes total graft occlusion that prevents blood flow through the graft to the revascularized part of the heart.
Bleeding | From the first procedure until one year after the second procedure
  Bleeding is assessed using the Bleeding Academic Research Consortium (BARC) classification, Thrombolysis In Myocardial Infarction (TIMI) bleeding classification and Global Use of Strategies to Open Occluded Coronary Arteries (GUSTO). classification
  BARC is subdivided into type zero (no bleeding) until five (probable/definite fatal bleeding), while the TIMI classification is divided into minimal, minor, and major. Gusto is subdivided into mild, moderate, and severe.
Quality of Life (QoL) using the Short-form 36 (SF-36) questionnaire | 14, 30, 90, 180 and 365 days after the second procedure
  QoL will be questioned with the Short-form 36 (SF-36) questionnaire.SF-36 scores range from 0 (worst) to 100 (best).
Quality of Life (QoL) using the Euro Quality of Life 5 dimensions (EQ-5D) questionnaire | 14, 30, 90, 180 and 365 days after the second procedure
  The Euro Quality of Life 5 dimensions (EQ-5D) questionnaire will be used to assess Quality of Life. Questions of the descriptive system are scored from one (no problem to perform activity) to five (severe problem/unable to perform activity). The scores are combined in order to calculate an index value (ranging from 0-1) that reflects the health state with one being the best health state. Moreover, the visual analogue scale ranges from 0 to 100 with 0 representing the worst health state and 100 the best health state.
Quality of Life (QoL) using the Seattle Angina Questionnaire short-form (SAQ-7) | 14, 30, 90, 180 and 365 days after the second procedure
  QoL will be questioned with the Seattle Angina Questionnaire short-form (SAQ-7). The overall summary score ranges from 0 to 100 where higher ratings indicate a better health state.
Quality of Life (QoL) using the Rose Dyspnea Scale (RDS) | 14, 30, 90, 180 and 365 days after the second procedure
  The Rose Dyspnea Scale (RDS) will be used to assess Quality of Life. RDS is scored between zero and four. Zero corresponds to no dyspnea with activity and four to dyspnea that severly limits activity.

CONTACTS AND LOCATIONS:
Overall Officials: Yoann Bataille, PhD, Principal Investigator — Jessa Hospital
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No